CLINICAL TRIAL: NCT04399551
Title: A Phase IIIb, Open-label, Hybrid Type III Trial Evaluating Implementation Strategies for Long-acting Cabotegravir Plus Long-acting Rilpivirine Every Two Months in HIV-1 Infected, Virologically Suppressed Adults in Select European Healthcare Settings
Brief Title: A Study Evaluating Implementation Strategies for Cabotegravir (CAB)+ Rilpivirine (RPV) Long-acting (LA) Injectables for Human Immunodeficiency Virus (HIV)-1 Treatment in European Countries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 213199
Record Dates: First submitted 2020-05-18; First posted 2020-05-22 (Actual); Results first posted 2023-05-19 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: HIV Infections
Keywords: Cabotegravir; Rilpivirine; Long-acting injectables; Patient study participants; Staff study participants
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Masking Description: This is an open-label study hence no blinding is required
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with HIV infection (Experimental): HIV-infected participants will receive CAB LA + RPV LA regimen for a month of oral lead in (OLI) at Day 1 followed by CAB LA + RPV LA injections at Months 1 and 2 and every 2 months (Q2M) thereafter.
  Interventions: Drug: CAB OLI; Drug: CAB LA; Drug: RPV OLI; Drug: RPV LA
- Staff study participants (SSP) (Other): Staff study participants will be randomized to receive standard implementation support (Arm-S; through visit(s) with the medication lead in their country, education on the medication, and patient and staff education/support materials) or through enhanced implementation support (Arm-E; through the addition of continuous quality improvement during the study).
  Interventions: Other: Continuous Quality Improvement (CQI) calls

INTERVENTIONS:
Drug: CAB OLI — CAB will be available as 30 milligrams (mg) tablet. It will be administered as one tablet once daily with food from Day 1 to Month 1.
  Arms: Participants with HIV infection
Drug: CAB LA — CAB LA 600 mg will be administered as intramuscular (IM) injection.
  Arms: Participants with HIV infection
Drug: RPV OLI — RPV will be available as 25 mg tablet. It will be administered as one tablet once daily with food from Day 1 to Month 1.
  Arms: Participants with HIV infection
Drug: RPV LA — RPV LA 900 mg will be administered as IM injection.
  Arms: Participants with HIV infection
Other: Continuous Quality Improvement (CQI) calls — CQI will be attended by the enhanced arm (Arm-E). The CQI calls will be conducted to identify problems/challenges, generate plans to address the challenges, and identify how to measure the change that results from the plan.
  Arms: Staff study participants (SSP)

SUMMARY:
The overall objective of the CAB LA + RPV LA clinical development program is to develop a highly effective, well-tolerated, two-drug, LA injectable regimen which has the potential to offer improved treatment convenience, compliance and improved quality of life for people living with HIV compared to current standard of care. This interventional study will examine different implementation strategies in different clinic settings across European countries to identify strategies which best meet the needs in each local context and involve both participants receiving study treatment CAB LA + RPV LA (patient study participants [PSP]) as well as the healthcare providers at the investigator site level (staff study participants [SSP]). SSPs consists of 2 groups: standard and enhanced arm.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older at the time of signing the informed consent.
* HIV-1 infected and must be suppressed on a guideline recommended active Highly active antiretroviral therapy (HAART) regimen for at least 6 months prior to screening. Any prior switch, defined as a change of a single drug or multiple drugs simultaneously, must have occurred due to tolerability/safety, access to medications, or convenience/simplification, and must not have been done for virologic failure (on treatment HIV-1 RNA more than or equal to [>=]200 c/mL).
* Documented evidence of at least two plasma HIV-1 RNA measurements <50 c/mL in the 12 months prior to Screening: at least one <6 months prior to screening and one 6-12 months prior to screening.
* Plasma HIV-1 RNA <50 c/mL at screening.
* A female participant is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG] test at screen and at Day 1), not lactating, and at least one of the following conditions applies:

  1. Non-reproductive potential is defined as:

     Pre-menopausal females with one of the following:
     * Documented tubal ligation.
     * Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion.
     * Hysterectomy.
     * Documented Bilateral Oophorectomy.
     * Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
  2. Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication, throughout the study, and for at least 30 days after discontinuation of all oral study medications and for at least 52 weeks after discontinuation of CAB LA and RPV LA.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and in this protocol. Eligible participants or their legal guardians (and next of kin when locally required), must sign a written informed consent form before any protocol-specified assessments are conducted. Enrolment of participants who are unable to provide direct informed consent is optional and will be based on local legal/regulatory requirements and site feasibility to conduct protocol procedures.
* French participants: In France, a participant will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion criteria:

* Within 6 months prior to screening, plasma HIV-1 RNA measurement >=50 c/mL.
* During the previous 12 months, any confirmed HIV-1 RNA measurement >=200 c/mL.
* Women who are pregnant, breastfeeding, or plan to become pregnant or breastfeed during the study.
* Any evidence of a current Center for Disease Control and Prevention (CDC) Stage 3 disease [CDC, 2014], except cutaneous Kaposi's sarcoma not requiring systemic therapy, and historical or current Cluster of Differentiation 4 (CD4)+ counts <200 cells per millimeter cube (cells/mm^3) are not exclusionary.
* Any pre-existing physical or mental condition (including substance use disorder) which, in the opinion of the investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
* Participants determined by the investigator to have a high risk of seizures, including participants with an unstable or poorly controlled seizure disorder. A participant with a prior history of seizure may be considered for enrolment if the investigator believes the risk of seizure recurrence is low.
* Participants who, in the investigator's judgment, pose a significant suicide risk. Participant's recent history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk.
* The participant has a tattoo, gluteal implant/ enhancements or other dermatological condition overlying the gluteus region which may interfere with interpretation of injection site reactions.
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antibody (anti-HBs) and HBV Deoxyribonucleic acid (DNA) as follows:

  * Participants positive for HBsAg are excluded.
  * Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded.
* Participants who are anticipated to require Hepatitis C virus (HCV) treatment within 12 months must be excluded. Asymptomatic individuals with chronic HCV infection will not be excluded; investigators must carefully assess if therapy specific for HCV infection is required. (HCV treatment on study may be permitted, following consultation and approval of the DAA based therapy being considered with the medical monitor).
* Participants with HCV co-infection will be allowed entry into this study if:

  1. Liver enzymes meet entry criteria.
  2. HCV disease has undergone appropriate work-up, and is not advanced. Additional information (where available) on participants with HCV coinfection at screening should include results from any liver biopsy, Fibroscan, ultrasound, or other fibrosis evaluation, history of cirrhosis or other decompensated liver disease, prior treatment, and timing/plan for HCV treatment.
  3. In the event that recent biopsy or imaging data is not available or inconclusive, the Fib-4 score will be used to verify eligibility:

     * Fib-4 score more than (>)3.25 is exclusionary.
     * Fib-4 score 1.45-3.25 requires Medical Monitor consultation Fibrosis 4 score formula:

(Age times Aspartate aminotransferase [AST]) / (Platelets times (square [Alanine aminotransferase]{ALT}).

* Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice or cirrhosis), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* History of liver cirrhosis with or without hepatitis viral co-infection.
* Ongoing or clinically relevant pancreatitis.
* Clinically significant cardiovascular disease, as defined by history/evidence of congestive heart failure, symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the participant prior to inclusion.
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to receive study medication.
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class. Current or anticipated need for chronic anti-coagulation with the exception of the use of low dose acetylsalicylic acid (less than or equal to [<=]325 mg per day) or hereditary coagulation and platelet disorders such as hemophilia or Von Willebrand Disease
* Any evidence of primary resistance based on the presence of any major known Integrase inhibitor (INI) or Non-nucleoside reverse transcriptase inhibitor (NNRTI) resistance-associated mutation, except for K103N, by any historical resistance test result.
* ALT >=5 times the upper limit of normal (ULN) or ALT >=3 times ULN and bilirubin >=1.5 times ULN (with >35 percent [%] direct bilirubin).
* Any verified Grade 4 laboratory abnormality. A single repeat test is allowed during the Screening phase to verify a result.
* Participant has estimated creatinine clearance <50 milliliters per minute (mL/min)/1.73 m^2 via the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to Day 1 of this study.
* Treatment with any of the following agents within 28 days of Day 1:

  * Radiation therapy.
  * Cytotoxic chemotherapeutic agents.
  * Tuberculosis therapy except for isoniazid (isonicotinylhydrazid [INH]).
  * Anti-coagulation agents.
  * Immunomodulators that alter immune responses such as chronic systemic corticosteroids, interleukins, or interferons.
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of screening.
* Use of medications which are associated with Torsade de Pointes must be discussed with the Medical Monitor to determine eligibility.
* Participants receiving any prohibited medication and who are unwilling or unable to switch to an alternate medication.
* A participant with known or suspected active Coronavirus Disease 2019 (COVID-19) infection OR contact with an individual with known COVID-19, within 14 days of study enrollment (World Health Organization [WHO] definitions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2023-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (15):
- Belgium (3):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
- France (4):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (2):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Utrecht
- Spain (4):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Cartagena (Murcia)
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Jonsson-Oldenbuttel C, Ghosn J, van der Valk M, Florence E, Vera F, De Wit S, Rami A, Bonnet F, Hocqueloux L, Hove K, Ait-Khaled M, DeMoor R, Bontempo G, Latham CL, Gutner CA, Iyer S, Gill M, Czarnogorski M, D'Amico R, van Wyk J. Safety and Effectiveness From the Cabotegravir and Rilpivirine Implementation Study in European Locations Study: Phase 3b Hybrid Type III Implementation Study Integrating Cabotegravir + Rilpivirine Long-Acting Into European Clinical Settings. J Acquir Immune Defic Syndr. 2024 Aug 15;96(5):472-480. doi: 10.1097/QAI.0000000000003448. Epub 2024 Jul 9. PMID 38985445
- [Derived] Gutner CA, Hocqueloux L, Jonsson-Oldenbuttel C, Vandekerckhove L, van Welzen BJ, Slama L, Crusells-Canales M, Sierra JO, DeMoor R, Scherzer J, Ait-Khaled M, Bontempo G, Gill M, Patel N, D'Amico R, Hove K, Baugh B, Barnes N, Hadi M, Low EL, Anand SB, Hamilton A, Garges HP, Czarnogorski M. Implementation of long-acting cabotegravir and rilpivirine: primary results from the perspective of staff study participants in the Cabotegravir And Rilpivirine Implementation Study in European Locations. J Int AIDS Soc. 2024 Jul;27(7):e26243. doi: 10.1002/jia2.26243. PMID 38978405

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 437 patient study participants (PSPs) [people living with HIV] were enrolled. 430 PSP received study treatment and were included in the safety population. Staff Study Participants (SSP) (HIV care providers, nurses/staff performing injections administrators/clinic managers) were not counted as enrolled. SSP were randomized based on implementation strategy - Enhanced (Arm-E) and Standard (Arm -S).
Pre-assignment Details: SSP provided input through surveys, semi-structured interviews and a selected group from the enhanced arm (Arm-E) participated in facilitation calls. Participant flow, Baseline characteristics or adverse events for SSP were not collected as it was not required per study design.
Groups:
- Patient Study Participants: PSPs received one tablet of cabotegravir (CAB) 30 milligrams (mg) + rilpivirine (RPV) 25 mg once daily from Day 1 for 1 month during the oral lead-in phase (OLI). Participants received last dose of oral regimen followed by CAB long-acting injectable (LA) 600 mg + RPV LA 900 mg injections in Month 1, one month later (Month 2), and every 2 months (Q2M) thereafter via intramuscular (IM) route.
Period: Overall Study
Arm/Group | Patient Study Participants
Started (Participants who received study treatment.) | 430
Completed | 402
Not Completed | 28
Not completed — Adverse Event | 15
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 3
Not completed — Lost to Follow-up | 2
Not completed — Protocol Deviation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 430
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.2 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 315
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 7
  Asian | 9
  Black Or African American | 76
  White | 336
  Multiple | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Acceptability of Implementation Measure (AIM-Imp) Score in SSP at Month 12
Description: The AIM-Imp was designed to assess the acceptability of an implementation process (i.e., perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory). The measure consists of four items/statements (1. The implementation support thus far meets my approval 2. The implementation support thus far is appealing to me 3. I like the implementation support I have received 4. I welcome implementation support for the CAB + RPV injection treatment), each with a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least acceptability and 5 the most acceptability.
Time Frame: Baseline (Month 1) and Month 12
Population: Full analysis set included all staff study participants (SSPs) who completed at least one survey at any timepoint. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Staff Study Participants - Enhanced Implementation Arm: SSPs included HIV care providers (HCPs), nurses/staff performing CAB + RPV LA injections, and administrators/clinic managers at each investigational site. They provided input using surveys, semi structured interviews (SSI) and via monthly facilitation calls. SSPs did not receive oral lead-in medication or CAB+RPV LA injections. This arm contains components like investigator meeting, SWAT meeting with sponsor team and principal clinic stakeholders, on-demand SWAT meeting, monthly continuous quality improvement (CQI) calls, face-to-face injection training, monthly FRAME assessment, access to patient and HCP level toolkit and CAB + RPV medical lead site visit.
- Staff Study Participants - Standard Implementation Arm: SSPs included HIV care providers (HCPs), nurses/staff performing CAB + RPV LA injections, and administrators/clinic managers at each investigational site. They provided input using surveys, semi structured interviews (SSI). SSPs did not receive oral lead-in medication or CAB+RPV LA injections. This arm contains components like investigator meeting, CAB + RPV medical lead site visit, access to patient and HCP level toolkit, virtual injection training and monthly FRAME assessment.
Arm/Group | Staff Study Participants - Enhanced Implementation Arm | Staff Study Participants - Standard Implementation Arm
Number analyzed (Participants) | 34 | 36
Scores on a scale
  Baseline (Month 1) | 3.8 (0.76) | 3.9 (0.75)
  Month 12: number analyzed (Participants) | 29 | 31
  Month 12 | 0.28 (0.828) | 0.33 (0.666)

2. Primary Outcome: Change From Baseline in Implementation Appropriateness Measure (IAM-Imp) Score in SSPs at Month 12
Description: The IAM-Imp is designed to assess the appropriateness of an implementation process (i.e., the perceived fit, relevance, or compatibility of the innovation for a given practice setting, provider, or consumer, and the perceived fit of the innovation to address a particular issue or problem). The IAM-Imp is a four-item/statement measure (1. The implementation support thus far seems fitting 2. The implementation support seems suitable for using the CAB + RPV injection treatment 3. The implementation support seems applicable for the CAB + RPV injection treatment 4. The implementation support seems like a good match) with a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least appropriateness and 5 the most appropriateness.
Time Frame: Baseline (Month 1) and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Staff Study Participants-Enhanced Implementation Arm: SSPs included HIV care providers (HCPs), nurses/staff performing CAB + RPV LA injections, and administrators/clinic managers at each investigational site. They provided input using surveys, semi structured interviews (SSI) and via monthly facilitation calls. SSPs did not receive oral lead-in medication or CAB+RPV LA injections. This arm contains components like investigator meeting, SWAT meeting with sponsor team and principal clinic stakeholders, on-demand SWAT meeting, monthly continuous quality improvement (CQI) calls, face-to-face injection training, monthly FRAME assessment, access to patient and HCP level toolkit and CAB + RPV medical lead site visit.
Arm/Group | Staff Study Participants-Enhanced Implementation Arm | Staff Study Participants - Standard Implementation Arm
Number analyzed (Participants) | 34 | 36
Scores on a scale
  Baseline (Month 1) | 3.8 (0.78) | 3.9 (0.78)
  Month 12: number analyzed (Participants) | 29 | 31
  Month 12 | 0.22 (0.740) | 0.31 (0.729)

3. Primary Outcome: Change From Baseline in Feasibility of Implementation Measure (FIM-Imp) Score at Month 12
Description: The FIM-Imp was a four-item/statement measure (1. The implementation support seems implementable in our clinic/practice 2. The implementation support seems possible in our clinic/practice 3. The implementation support seems doable in our clinic/practice 4. The implementation support seems easy to use in our clinic/practice) and was measured on a five-point rating scale (1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, and 5 = completely agree). The mean score ranges from 1 to 5 with 1 indicating the least feasibility and 5 the most feasibility.
Time Frame: Baseline (Month 1) and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Staff Study Participants - Enhanced Implementation Arm | Staff Study Participants - Standard Implementation Arm
Number analyzed (Participants) | 34 | 36
Scores on a scale
  Baseline (Month 1) | 4.0 (0.66) | 4.0 (0.64)
  Month 12: number analyzed (Participants) | 29 | 31
  Month 12 | 0.06 (1.047) | 0.34 (0.773)

4. Secondary Outcome: Number of Staff Study Participants That Discussed Facilitators for Acceptability Assessed Via Semi Structured Interviews (SSIs)
Description: A semi-structured interview guide was designed to support the discussion surrounding experience with the implementation of CAB+RPV LA injection treatment. The interview guide topics were informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework and Proctor Outcomes to facilitate discussions on the acceptability from the SSPs' perspective. The results for facilitators that are integral to successful implementation are presented.
Time Frame: Up to 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Study Participants - Standard Implementation Arm | Staff Study Participants - Enhanced Implementation Arm
Number analyzed (Participants) | 32 | 30
Participants
  Improved Patient's Quality of Life | 0 | 1
  Injection pain management | 2 | 0
  No commute to clinic | 1 | 3

5. Secondary Outcome: Number of Staff Study Participants That Discussed Barriers for Acceptability Assessed Via SSIs
Description: A semi-structured interview guide was designed to support the discussion surrounding experience with for the implementation of CAB+RPV LA injection treatment. The interview guide topics were informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework and Proctor Outcomes to facilitate discussions on the acceptability from the SSPs' perspective. The results for barriers that are integral to successful implementation are presented.
Time Frame: Up to 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Study Participants - Standard Implementation Arm | Staff Study Participants - Enhanced Implementation Arm
Number analyzed (Participants) | 32 | 30
Participants | 1 | 1

6. Secondary Outcome: Number of Staff Study Participants That Discussed Facilitators for Appropriateness Assessed Via SSIs
Description: A semi-structured interview guide was designed to support the discussion surrounding experience with for the implementation of CAB+RPV LA injection treatment. The interview guide topics were informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework and Proctor Outcomes to facilitate discussions on the appropriateness from the SSPs' perspective. The results for facilitators that are integral to successful implementation are presented.
Time Frame: Up to 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Study Participants - Standard Implementation Arm | Staff Study Participants - Enhanced Implementation Arm
Number analyzed (Participants) | 32 | 30
Participants
  Patient characteristics | 1 | 2
  Patient selection | 0 | 2
  Hours of home visit | 1 | 1

7. Secondary Outcome: Number of Staff Study Participants That Discussed Barriers for Appropriateness Assessed Via SSIs
Description: A semi-structured interview guide was designed to support the discussion surrounding experience with for the implementation of CAB+RPV LA injection treatment. The interview guide topics were informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework and Proctor Outcomes to facilitate discussions on the appropriateness from the SSPs' perspective. The results for barriers that are integral to successful implementation are presented.
Time Frame: Up to 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Study Participants - Standard Implementation Arm | Staff Study Participants - Enhanced Implementation Arm
Number analyzed (Participants) | 32 | 30
Participants | 0 | 0

8. Secondary Outcome: Number of Staff Study Participants That Discussed Facilitators for Feasibility Assessed Via SSIs
Description: A semi-structured interview guide was designed to support the discussion surrounding experience with for the implementation of CAB+RPV LA injection treatment. The interview guide topics were informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework and Proctor Outcomes to facilitate discussions on the feasibility from the SSPs' perspective. The results for facilitators that are integral to successful implementation are presented.
Time Frame: Up to 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Study Participants - Standard Implementation Arm | Staff Study Participants - Enhanced Implementation Arm
Number analyzed (Participants) | 32 | 30
Participants
  Clinic or unit characteristics (e.g., autonomy, size, flexibility) | 2 | 3
  Experience with the medication | 0 | 1
  Implementation processes | 2 | 2
  Medication storage | 2 | 1
  Number of patients | 1 | 2
  Nursing staff in consultation department | 0 | 1
  Pharmacy flexibility | 0 | 1
  Room/space characteristics | 1 | 1
  Staff availability | 0 | 2
  Staff characteristics (e.g., experience, qualification, motivation) | 6 | 8
  Training | 1 | 0
  ViiV support and materials | 3 | 1

9. Secondary Outcome: Number of Staff Study Participants That Discussed Barriers for Feasibility Assessed Via SSIs
Description: A semi-structured interview guide was designed to support the discussion surrounding experience with for the implementation of CAB+RPV LA injection treatment. The interview guide topics were informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework and Proctor Outcomes to facilitate discussions on the feasibility from the SSPs' perspective. The results for barriers that are integral to successful implementation are presented.
Time Frame: Up to 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Study Participants - Standard Implementation Arm | Staff Study Participants - Enhanced Implementation Arm
Number analyzed (Participants) | 32 | 30
Participants | 0 | 0

10. Secondary Outcome: Change From Baseline in Implementation Leadership Scale (ILS) Score at Month 12
Description: The ILS is a 12-item (facilitate implementation, obstacles, clear department standards, knowledge, ability to answer questions, awareness of concept, recognition, support employee efforts to learn, support employee efforts to use intervention, persevere(s) through the ups and downs, carries on through the challenges and reaction to criticial issues) measure that assesses SSP understanding of the degree to which leadership in their clinic/practice setting is proactive, knowledgeable, supportive, and perseverant with regards to implementing the CAB LA + RPV LA injection treatment in their settings. The items are measured on a five-point rating scale (1 = very great extent, 2 = great extent, 3 = moderate extent, 4 = slight extent, and 5 = not at all). The mean score ranges from 1 to 5. Higher the score means less understanding in leadership.
Time Frame: Baseline (Month 1) and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Staff Study Participants - Enhanced Implementation Arm | Staff Study Participants - Standard Implementation Arm
Number analyzed (Participants) | 34 | 35
Scores on a scale
  Baseline (Month 1) | 2.3 (0.86) | 2.0 (0.81)
  Month 12: number analyzed (Participants) | 30 | 31
  Month 12 | -0.1 (1.19) | 0.2 (0.51)

11. Secondary Outcome: Absolute Values of Implementation Climate Scale (ICS) Scores at Month 1 and Month 12
Description: The ICS is a 9 item (team's main goals, importance of implementation, top priority, workshops, treatment training, training material, staff adaptability, flexibility, openness to new intervention) measure that assesses SSPs' perceptions of their team (i.e., the people that they work with) while using the CAB LA + RPV LA injection treatment in their clinic/practice setting. The items were measured on a five-point rating scale (1 = very great extent, 2 = great extent, 3 = moderate extent, 4 = slight extent, and 5 = not at all). The mean score ranges from 1 to 5. Higher the score means less seriousness for implementation in staff.
Time Frame: Month 1 and Month 12
Population: Full Analysis Set. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Staff Study Participants - Enhanced Implementation Arm: SSPs included HIV care providers (HCPs), nurses/staff performing CAB + RPV LA injections, and administrators/clinic managers at each investigational site. They provided input using surveys, semi structured interviews (SSI) and via monthly facilitation calls. SSPs did not receive oral lead-in medication or CAB+RPV LA injections. This arm contains components like investigator meeting, SWAT meeting with sponsor team and principle clinic stakeholders, on-demand SWAT meeting, monthly continuous quality improvement (CQI) calls, face-to-face injection training, monthly FRAME assessment, access to patient and HCP level toolkit and CAB + RPV medical lead site visit.
Arm/Group | Staff Study Participants - Enhanced Implementation Arm | Staff Study Participants - Standard Implementation Arm
Number analyzed (Participants) | 34 | 35
Scores on a scale
  Month 1 | 2.5 (0.65) | 2.8 (0.80)
  Month 12: number analyzed (Participants) | 30 | 31
  Month 12 | 2.7 (0.72) | 2.6 (0.80)

12. Secondary Outcome: Number of Modifications Reported by SSPs Assessed Via FRAME-IS
Description: The Framework for Reporting Adaptations and Modifications to Evidence-based interventions - Implementation Strategies (FRAME-IS) was a seven-question measure (contained both open and closed categorical questions) used to record details the modifications made to the implementation of the CAB LA + RPV LA injection treatment procedures.
Time Frame: Month 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
Population: as for outcome 1
Measure: Number; unit: Number of Modifications
Arm/Group | Staff Study Participants - Enhanced Implementation Arm | Staff Study Participants - Standard Implementation Arm
Number analyzed (Participants) | 34 | 35
Number of Modifications
  Month 2 | 15 | 7
  Month 3 | 10 | 2
  Month 4 | 5 | 2
  Month 5 | 1 | 1
  Month 6 | 3 | 0
  Month 7 | 4 | 0
  Month 8 | 0 | 0
  Month 9 | 3 | 0
  Month 10 | 0 | 0
  Month 11 | 3 | 1
  Month 12 | 0 | 1

13. Secondary Outcome: Number of Plan, Do, Study, Act (PDSA) Cycles Developed During the Continuous Quality Improvement (CQI) Calls Course
Description: CQI were a 60 minutes calls involved working through a plan to address the identified barriers, optimize processes, and evaluate these efforts. This process of addressing barriers was guided by a series of Plan, Do, Study, Act (PDSA) cycles. Number of PDSA cycles developed are presented.
Time Frame: Month 2 to Month 7
Population: Full Analysis Set. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Cycles
Groups:
- Staff Study Participants (SSP): SSPs included HIV care providers (HCPs), nurses/staff performing CAB + RPV LA injections, and administrators/clinic managers at each investigational site. They provided input through the use of surveys, semi structured interviews (SSI) and via monthly facilitation calls. SSPs did not receive oral lead-in medication or CAB+RPV LA injections.
Arm/Group | Staff Study Participants (SSP)
Number analyzed (Participants) | 18
Cycles | 23

14. Secondary Outcome: Number of Participants Spending Average Time in the Clinic/Practice for Each Injection Visit Assessed Via Questionnaire
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question. The average time was categorized as: Up to 20 Minutes, Up to 40 Minutes, Up to 60 Minutes, Up to 90 Minutes, More than 90 Minutes and missing. Missing include participants who did not provide a response for the question.
Time Frame: Up to Month 12
Population: Patient study participants (PSPs) included all participants who successfully completed the survey at Month 12. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Up to 20 Minutes | 71
  Up to 40 Minutes | 134
  Up to 60 Minutes | 99
  Up to 90 Minutes | 48
  More than 90 Minutes | 19
  Missing | 8

15. Secondary Outcome: Number of Participants Spending Average Time in an Exam Room Waiting for a Nurse (or Other Healthcare Provider) to Get the Injection Administered Assessed Via Questionnaire
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question. The average time was categorized as: Up to 10 Minutes, 11-20 Minutes, 21-30 Minutes, 31-45 Minutes, More than 45 Minutes and Missing. Missing include participants who did not provide a response for the question.
Time Frame: Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Up to 10 Minutes | 190
  11-20 Minutes | 100
  21-30 Minutes | 54
  31-45 Minutes | 25
  More than 45 Minutes | 5
  Missing | 5

16. Secondary Outcome: Number of Participants Rating Acceptability With the Amount of Time Spent in The Clinic/Practice for Each Injection Visit Assessed Via Questionnaire
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question. The rating of acceptability was categorized as extremely acceptable, very acceptable, somewhat acceptable, a little acceptable, not at all acceptable and missing. Missing include participants who did not provide a response for the question.
Time Frame: Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Extremely acceptable | 140
  Very acceptable | 151
  Somewhat acceptable | 72
  A little acceptable | 11
  Not at all acceptable | 0
  Missing | 5

17. Secondary Outcome: Number of Participants Rating Acceptability to Come to the Clinic/Practice Every 2 Months for the Injection Visit Assessed Via Questionnaire
Description: as for outcome 16
Time Frame: Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Extremely acceptable | 163
  Very acceptable | 154
  Somewhat acceptable | 51
  A little acceptable | 6
  Not at all acceptable | 0
  Missing | 5

18. Secondary Outcome: Number of Participants Taking Time Off From Work to Attend Appointment Assessed Via Questionnaire
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question. The time off responses were categorized as Whole day annual leave, Half day annual leave, Whole day sick leave, Half day sick leave, Whole day unpaid, Half day unpaid, Other, Not taken time off and missing. Missing include participants who did not provide a response for the question.
Time Frame: Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Whole day annual leave | 27
  Half day annual leave | 20
  Whole day sick leave | 5
  Half day sick leave | 3
  Whole day unpaid | 9
  Half day unpaid | 20
  Other | 64
  Not taken Time Off | 222
  Missing | 9

19. Secondary Outcome: Number of Participants With Time it Took Them to Get to the Clinic Where They Receive HIV Treatment/Check-ups Assessed Via Questionnaire
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question. The responses were categorized as Up to 15 minutes, 16-30 minutes, 31-45 minutes, 46-60 minutes, More than 60 minutes, and missing. Missing include participants who did not provide a response for the question.
Time Frame: Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Up to 15 minutes | 66
  16-30 minutes | 138
  31-45 minutes | 87
  46-60 minutes | 44
  More than 60 minutes | 39
  Missing | 5

20. Secondary Outcome: Number of Participants Who Seek Additional Care From a Dependent to Attend Appointment Assessed Via Questionnaire
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question. The responses were categorized as Yes, No, Not Applicable and Missing. Missing include participants who did not provide a response for the question.
Time Frame: Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Yes | 16
  No | 318
  Not Applicable | 39
  Missing | 6

21. Secondary Outcome: Number of Participants That Endorsed Type of Transportation Used to Attend Appointments
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question. The responses were categorized as Taxi- Transportation service, Dropped-off, Private vehicle, Bicycle/scooter/ skateboard/ walked, Public transport and Missing. Missing include participants who did not provide a response for the question.
Time Frame: Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Taxi-Transportation service | 13
  Dropped-off | 12
  Private vehicle | 164
  Bicycle/ scooter/ skateboard/ walked | 49
  Public transport | 138
  Missing | 3

22. Secondary Outcome: Number of Participants Taking Time Off From Work to Recover From Any Injection Site Reaction Issue Assessed Via Questionnaire
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question. The time off responses were categorized as No, Yes - On the day of receiving the treatment, Yes - One day after receiving the treatment, Yes-Two days after receiving the treatment, Yes-More than two days after receiving the treatment, Not Applicable, Missing and Missing Response for 'Yes'. Missing include participants who did not provide a response for the question. Missing Response for 'Yes' include participants who responded 'Yes' but did not provide duration of time off.
Time Frame: Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  No | 294
  Yes, on the day of receiving the treatment | 45
  Yes, one day after receiving the treatment | 9
  Yes, two days after receiving the treatment | 7
  Yes, more than two days after receiving the treatment | 5
  Not Applicable | 16
  Missing | 5
  Missing response for 'Yes' | 2

23. Secondary Outcome: Number of Participants Rating Convenience of Clinic/Practice's Procedures for Scheduling Injections Assessed Via Questionnaire
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question. The convenience responses were categorized as Extremely convenient, Very convenient, Somewhat convenient, A little convenient, Not at all convenient, and Missing. Missing include participants who did not provide a response for the question.
Time Frame: Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Extremely convenient | 175
  Very convenient | 154
  Somewhat convenient | 43
  A little convenient | 4
  Not at all convenient | 0
  Missing | 3

24. Secondary Outcome: Number of Participants Rating Convenience of Clinic/Practice's Procedures for Rescheduling Injections Assessed Via Questionnaire
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question. The responses were categorized as Extremely convenient, Very convenient, Somewhat convenient, A little convenient, Not at all convenient, Not applicable; I did not have to reschedule and Missing. Missing include participants who did not provide a response for the question.
Time Frame: Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Extremely convenient | 158
  Very convenient | 153
  Somewhat convenient | 25
  A little convenient | 2
  Not at all convenient | 0
  Not applicable; I did not have to schedule | 39
  Missing | 2

25. Secondary Outcome: Number of Participants Rating Feelings About Getting CAB+RPV Injection Treatment Assessed Via Questionnaire
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question. The responses were categorized as Extremely positive, Very positive, Somewhat positive, A little positive, Not at all positive and Missing. Missing include participants who did not provide a response for the question.
Time Frame: Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Extremely positive | 234
  Very positive | 112
  Somewhat positive | 23
  A little positive | 4
  Not at all positive | 0
  Missing | 6

26. Secondary Outcome: Number of Participants That Rated Perceived Knowledge About CAB+RPV Injection Treatment Assessed Via Questionnaire
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question. The responses were categorized as Extremely knowledgeable, Very knowledgeable, Somewhat knowledgeable, A little knowledgeable, Not at all knowledgeable and Missing. Missing include participants who did not provide a response for the question.
Time Frame: Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Extremely knowledgeable | 124
  Very knowledgeable | 188
  Somewhat knowledgeable | 57
  A little knowledgeable | 6
  Not at all knowledgeable | 0
  Missing | 4

27. Secondary Outcome: Number of Participants With Appointment Reminders Received Assessed Via Questionnaire
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question.The responses were categorized as Phone calls, Text/SMS messages, Existing clinic app, E-mail, Reminder in the mail, Another reminder and I did not receive reminders. The responses are not mutually exclusive.
Time Frame: Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Phone calls | 80
  Text/SMS messages | 275
  Existing clinic app | 48
  E-mail | 161
  Reminder in the mail | 21
  Another reminder | 3
  I did not receive reminders | 14

28. Secondary Outcome: Number of Participants Who Rated Helpfulness of Appointment Outside of Typical Work Times Assessed Via Questionnaire
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question. The responses were categorized as Extremely helpful, Very helpful, Somewhat helpful, A Little helpful, Not at all helpful and Missing. Missing include participants who did not provide a response for the question.
Time Frame: Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Extremely helpful | 135
  Very helpful | 123
  Somewhat helpful | 50
  A Little helpful | 38
  Not at all helpful | 28
  Missing | 5

29. Secondary Outcome: Number of Participants That Rated Agreement in Recommending the CAB+RPV Injections to Others Assessed Via Questionnaire
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question. The responses were categorized as Completely agree, Agree, Neutral, Disagree, Completely disagree and Missing. Missing include participants who did not provide a response for the question.
Time Frame: Month 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Completely agree | 283
  Agree | 75
  Neutral | 15
  Disagree | 1
  Completely disagree | 1
  Missing | 4

30. Secondary Outcome: Number of Participants With Things Tried to Reduce Soreness Following Injections Assessed Via Questionnaire
Description: Study-specific questions were developed to gather data on the facilitators and barriers of the CAB LA + RPV LA injection treatment. The response options are different for each question. The responses were categorized as Take over-the-counter pain relievers, Use a hot compress, Use a cold compress, Avoid sitting for long periods of time, Light stretching and exercise, None of the above, Other and I don't get sore after my injections.
Time Frame: Month 12
Population: Patient study participants (PSPs) included all participants who successfully completed the survey at Month 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Take over-the-counter pain relievers | 139
  Use a hot compress | 20
  Use a cold compress | 19
  Avoid sitting for long periods of time | 87
  Light stretching and exercise | 71
  None of the above | 61
  Other | 31
  I don't get sore after my injections | 72

31. Secondary Outcome: Number of PSPs That Discussed Facilitators for Acceptability Assessed Via Semi Structured Interviews (SSIs)
Description: A semi-structured interview guide was developed to support the discussion surrounding experience with for the implementation of CAB+RPV LA injection treatment. The interview guide topics were informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework and Proctor Outcomes to facilitate discussions on the Acceptability, Appropriateness, Feasibility, and Sustainability from the PSPs' perspective. Results of number of PSPs that discussed facilitators for acceptability are presented.
Time Frame: Up to Month 12
Population: Patient study participants (PSPs) who participated in interviews were analysed. Only those participants with data available at the specified time points were analysed.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 110
Participants
  Feeling informed about CAB+RPV LA injection | 105
  Overall positive experience with CAB+RPV LA | 100
  Acceptable overall experience at clinic | 82
  In-person communication with HCP | 76
  Not thinking and/or worrying about taking medication | 66
  Experienced injector | 64
  Acceptable clinic hours to receive CAB+RPV LA injections | 51
  CAB+RPV LA injection experience met expectations | 43
  Patient travel facilitation | 33
  CAB+RPV LA injection experience better than expected | 32
  Staff responsiveness | 34
  Number of visits | 30
  Satisfaction with rescheduling process | 29
  Distance to clinic | 27
  Not being reminded about HIV | 26
  Acceptable time spent in clinic | 25
  Treatment adherence | 24
  Gaining a sense of freedom | 24
  Discreet treatment | 23
  Communication with staff | 22
  Reduced stigma due to CAB+RPV LA injection | 22
  Reduction in injection pain | 20
  [Patient-perspective] Medication for injection pain management | 19
  Reduced stress or worry due to CAB+RPV LA injection | 19
  HCP advice on pain management | 18
  [Patient-perspective] Activities to avoid for injection pain management | 16
  Website and/or internet | 15
  Characteristics of HCP communication | 14
  Written materials and brochures | 14
  Study materials | 14
  Time of informing | 13
  Medication collection, storage and/or preparation | 12
  Fewer side effects | 12
  Time-saving approach | 12
  [Patient-perspective] Activities to do for injection pain management | 11
  Administration in other clinical setting | 11

32. Secondary Outcome: Number of PSPs That Discussed Barriers for Acceptability Assessed Via SSIs
Description: A semi-structured interview guide was developed to support the discussion surrounding experience with for the implementation of CAB+RPV LA injection treatment. The interview guide topics were informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework and Proctor Outcomes to facilitate discussions on the Acceptability, Appropriateness, Feasibility, and Sustainability from the PSPs' perspective. Results of number of PSPs that discussed barriers for acceptability are presented.
Time Frame: Up to Month 12
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 110
Participants
  Injection side effects including pain (Topic - Treatment Components Difficult for PSP) | 67
  Injection side effects including pain (Topic-Experienced Challenges to Receive CAB+PRV LA Injection) | 33
  CAB+RPV LA injection experience worse than expected | 11
  Waiting time | 11

33. Secondary Outcome: Number of PSPs That Discussed Facilitators for Appropriateness Assessed Via SSIs
Description: A semi-structured interview guide was developed to support the discussion surrounding experience with for the implementation of CAB+RPV LA injection treatment. The interview guide topics were informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework and Proctor Outcomes to facilitate discussions on the Acceptability, Appropriateness, Feasibility, and Sustainability from the PSPs' perspective. Results of number of PSPs that discussed facilitators for appropriateness are presented.
Time Frame: Up to Month 12
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 110
Participants | 0

34. Secondary Outcome: Number of PSPs That Discussed Barriers for Appropriateness Assessed Via SSIs
Description: A semi-structured interview guide was developed to support the discussion surrounding experience with for the implementation of CAB+RPV LA injection treatment. The interview guide topics were informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework and Proctor Outcomes to facilitate discussions on the Acceptability, Appropriateness, Feasibility, and Sustainability from the PSPs' perspective. Results of number of PSPs with barriers for appropriateness are presented.
Time Frame: Up to Month 12
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 110
Participants
  Patient fearing or squeamish about injections | 22
  Patients not tolerating intramuscular injection | 12

35. Secondary Outcome: Number of PSPs That Discussed Facilitators for Feasibility Assessed Via SSIs
Description: A semi-structured interview guide was developed to support the discussion surrounding experience with for the implementation of CAB+RPV LA injection treatment. The interview guide topics were informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework and Proctor Outcomes to facilitate discussions on the Acceptability, Appropriateness, Feasibility, and Sustainability from the PSPs' perspective. Results of number of PSPs that discussed facilitators for feasibility are presented.
Time Frame: Up to Month 12
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 110
Participants
  Person to contact during CARISEL study | 102
  [Patient-perspective] Calendar, Diary, Notes and/or Reminders | 69
  No missed appointment and/or rescheduling | 65
  Target date explained | 57
  Easy to contact | 57
  Contacting clinic staff during CARISEL study | 52
  Home administration by HCP | 41
  No issues due to transportation and/or parking | 37
  No challenges to receive CAB+RPV LA injection | 33
  Not contacting clinic staff during CARISEL study | 31
  No issues due to work | 28
  Clinic Reminder [all types] | 27
  Term of target date helpful | 25
  [Patient-perspective] Setting reminders | 23
  CAB+RPV LA administration at GP office | 22
  CAB+RPV LA administration at nurse office and/or healthcare centers | 19
  No issues to attend visits due to childcare or family commitments | 16
  [Patient-perspective] Arrangements at work | 16
  Clinic reminder: Text and/or SMS | 14
  [Patient-perspective] Appointment scheduling strategies | 14
  No issues due to clinic hours | 13

36. Secondary Outcome: Number of PSPs That Discussed Barriers for Feasibility Assessed Via SSIs
Description: A semi-structured interview guide was developed to support the discussion surrounding experience with for the implementation of CAB+RPV LA injection treatment. The interview guide topics were informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework and Proctor Outcomes to facilitate discussions on the Acceptability, Appropriateness, Feasibility, and Sustainability from the PSPs' perspective. Results of number of PSPs that discussed barriers for feasibility are presented.
Time Frame: Up to Month 12
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 110
Participants
  Target date not explained | 38
  Missed appointment and/or rescheduling | 23
  Issues due to work | 21
  Issues due to transportation and/or parking | 14

37. Secondary Outcome: Change From Baseline in Acceptability of Intervention Measure (AIM) Score in PSPs at Month 12
Description: AIM assesses the acceptability of an intervention (i.e., perception among stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory). It is a four-item (1. The CAB+RPV injection treatment meets my approval for treating my HIV, 2. The CAB+RPV injection treatment is appealing to me, 3. I like the CAB+RPV injection treatment for my HIV, 4. I welcome the CAB+RPV injection treatment for my HIV) measure with a five-point rating scale, where 1=completely disagree, 2=disagree, 3=neither agree nor disagree, 4=agree, and 5=completely agree. The mean score ranges from 1 to 5 with 1 indicating the least acceptability and 5 the most acceptability.
Time Frame: Baseline (Month 1) and Month 12
Population: PSPs who completed the surveys at the relevant timepoints were included in the analysis. Only those participants with data available at the specified time points were analysed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 424
Scores on a scale
  Baseline (Month 1) | 4.55 (0.666)
  Month 12: number analyzed (Participants) | 377
  Month 12 | 0.10 (0.834)

38. Secondary Outcome: Change From Baseline in Intervention Appropriateness Measure (IAM) Score in PSPs at Month 12
Description: IAM assesses the appropriateness of an intervention (i.e., the perceived fit, relevance, or compatibility of the innovation for a given practice setting, provider, or consumer; and the perceived fit of the innovation to address a particular issue or problem). It is a four-item (1. The CAB+RPV injection treatment is fitting for my life, 2. The CAB+RPV injection treatment is suitable for my life, 3. The CAB+RPV injection treatment is applicable to my life, 4. The CAB+RPV injection treatment is a good match for my life) measure with a five-point rating scale, where 1=completely disagree, 2=disagree, 3=neither agree nor disagree, 4=agree, and 5=completely agree. The mean score ranges from 1 to 5 with 1 indicating the least appropriateness and 5 the most appropriateness.
Time Frame: Baseline (Month 1) and Month 12
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 423
Scores on a scale
  Baseline (Month 1) | 4.47 (0.762)
  Month 12: number analyzed (Participants) | 376
  Month 12 | 0.13 (0.928)

39. Secondary Outcome: Change From Baseline in Feasibility of Intervention Measure (FIM) Score in PSPs at Month 12
Description: The four-item (1. The CAB+RPV injection treatment seems implementable in my life 2. The CAB+RPV injection treatment every 2 months is possible for me to use 3. The CAB+RPV injection treatment every 2 months seems doable in my life 4. The CAB+RPV injection treatment every 2 months seems easy to use in my life). FIM assesses perceived intervention feasibility. The items are measured on a five-point rating scale, where 1=completely disagree, 2=disagree, 3=neither agree nor disagree, 4=agree, and 5=completely agree. The mean score ranges from 1 to 5 with 1 indicating the least feasibility and 5 the most feasibility.
Time Frame: Baseline (Month 1) and Month 12
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 424
Scores on a scale
  Baseline (Month 1) | 4.51 (0.672)
  Month 12: number analyzed (Participants) | 376
  Month 12 | 0.07 (0.857)

40. Secondary Outcome: Associated Person Clinical Sustainability Assessment Tool (APCSAT) Average Domain Score at Month 12
Description: The APCSAT is a 35-item measure that assesses SSP impressions of the data in their clinic. Sustainability refers to the ability to maintain and expand the CAB LA + RPV LA injection treatment and its benefits over time. SSPs were asked to rate their clinic/practice along a range of specific domains that affect sustainability, including: 'Engages Staff & Leadership,' 'Engaging Stakeholders,' 'Monitoring and Evaluation,' 'Implementation & Training,' 'Outcomes & Effectiveness,' 'Workflow Integration,' and 'Organizational Readiness.' Five items were presented to SSPs in each section. The items were measured on a seven-point rating scale (1 = little to no extent to 7 = to a very great extent. Domain total was divided by the total number of items with a score to get average score.
Time Frame: Month 12
Population: Full Analysis Set. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Staff Study Participants - Enhanced Implementation Arm | Staff Study Participants - Standard Implementation Arm
Number analyzed (Participants) | 32 | 30
Scores on a scale
  Engages Staff & Leadership | 5.57 (0.72) | 5.58 (0.49)
  Engaging Stakeholders | 5.00 (1.06) | 5.05 (0.79)
  Monitoring and Evaluation | 5.37 (0.16) | 5.49 (0.11)
  Implementation & Training | 5.62 (0.56) | 5.56 (0.43)
  Outcomes & Effectiveness | 5.39 (0.70) | 5.41 (0.69)
  Workflow Integration | 5.46 (0.35) | 5.23 (0.34)
  Organizational Readiness | 5.30 (0.32) | 5.05 (0.36)

41. Secondary Outcome: Percentage of PSP Receiving Injections Within Target Window
Description: The target window for participants to receive injection was from Day -7 to Day 7.
Time Frame: Day -7 to Day 7 of Month 2, 4, 6, 8, 10 and 12
Population: Safety population included all enrolled participants who received at least one dose of CAB + RPV Oral or CAB LA + RPV LA.
Measure: Number; unit: Percentage of Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 430
Percentage of Participants
  Month 2 | 99
  Month 4 | 93
  Month 6 | 91
  Month 8 | 91
  Month 10 | 94
  Month 12 | 91

42. Secondary Outcome: Percentage of PSPs With Plasma HIV-1 Ribonucleic Acid (RNA) Less Than (<)50 Copies Per Milliliter (c/ml)
Description: Plasma samples were collected from the participant at specific time points.
Time Frame: Month 1, 2, 4, 8 and 12
Population: Safety population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Patient Study Participants: Participants with HIV received one tablet of Cabotegravir (CAB) 30 milligrams (mg) + Rilpivirine (RPV) 25 mg once daily from Day 1 for 1 month during the oral lead-in phase (OLI). Participants received last dose of oral regimen followed by CAB long-acting injectable (LA) 600 mg + RPV LA 900 mg injections in Month 1, one month later (Month 2), and every 2 months (Q2M) thereafter via intramuscular (IM) route.
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 430
Percentage of Participants
  Month 1 | 99 [97.0 to 99.5]
  Month 2 | 96 [93.7 to 97.7]
  Month 4 | 93 [90.5 to 95.4]
  Month 8 | 86 [82.7 to 89.4]
  Month 12 | 87 [83.2 to 89.8]

43. Secondary Outcome: Number of Participants With Confirmed Virologic Failure (CVF) Over Time
Description: CVF was defined as rebound as indicated by two consecutive plasma HIV-1 RNA levels >=200 c/ml.
Time Frame: Month 1, 2, 4, 8, 10 and 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 430
Participants
  Month 1 | 0
  Month 2 | 0
  Month 4 | 0
  Month 6 | 0
  Month 8 | 0
  Month 10 | 1
  Month 12 | 0

44. Secondary Outcome: Number of PSPs With Adverse Events (AEs) And Serious AEs (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose may result in death or is life-threatening or requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity or is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment or is associated with liver injury and impaired liver function.
Time Frame: Up to 12 Months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 430
Participants
  Any AEs | 420
  Any SAEs | 15

45. Secondary Outcome: Number of PSPs Discontinuing Treatment Due to AEs
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 12 Months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 430
Participants | 2

46. Secondary Outcome: Number of PSP With Preference for Therapy Assessed Via Preference Questionnaire
Description: PSPs were asked to think about their experience of using the long-acting injectable medication versus the daily oral HIV medication, and to select their preferred treatment and all the reasons that support their preference. Results are categorized as: 'long-acting injectable HIV medication', 'daily oral HIV medication', 'no preference', Missing and Erroneous. Missing include participants who did not provide a response for the question. PSPs who completed this question incorrectly (i.e., checked reasons without a ticking a leading preference or checked more than one leading preference box) were included in Erroneous.
Time Frame: Up to 12 Months
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Study Participants
Number analyzed (Participants) | 379
Participants
  Daily oral HIV medication | 2
  Long-acting injectable HIV medication | 275
  No preference | 0
  Missing | 2
  Erroneous | 100

47. Primary Outcome: Number of Participants That Discussed Themes Arising Out of Qualitative Semi-structured Interviews Which Are Coded as Acceptability
Description: A semi-structured interview guide was designed to support the discussion surrounding experience with the implementation of CAB+RPV LA injection treatment. The interview guide topics were informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework and Proctor Outcomes to facilitate discussions on the acceptability from the SSPs' perspective. The results of themes that are integral to successful implementation are presented based on implementation strategies.
Time Frame: Up to 12 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Study Participants - Standard Implementation Arm | Staff Study Participants - Enhanced Implementation Arm
Number analyzed (Participants) | 32 | 30
Participants
  Positive opinion about CAB+RPV LA | 28 | 28
  Negative opinion about CAB+RPV LA | 0 | 0
  Ambivalent opinion about CAB+RPV LA | 3 | 1
  Opinion about CAB+RPV LA did not change | 15 | 14
  Opinion about CAB+RPV LA changed | 9 | 11
  Treatment and/or its implementation is better than expected | 7 | 11
  Treatment and/or its implementation is worse than expected | 2 | 0
  Implementation facilitators reported | 16 | 19
  Did NOT encounter resistance to using CAB+RPV LA | 8 | 19
  ADMINISTRATION OUTSIDE CLINIC: Other clinical settings | 15 | 15
  ADMINISTRATION OUTSIDE CLINIC: Self-administered | 20 | 23
  What would do differently | 2 | 4

48. Primary Outcome: Number of Participants That Discussed Themes Arising Out of Qualitative Semi-structured Interviews Which Are Coded as Appropriateness
Description: A semi-structured interview guide was designed to support the discussion surrounding experience with the implementation of CAB+RPV LA injection treatment. The interview guide topics were informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework and Proctor Outcomes to facilitate discussions on the appropriateness from the SSPs' perspective. The results of themes that are integral to successful implementation are presented based on implementation strategies.
Time Frame: Up to Month 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Study Participants - Standard Implementation Arm | Staff Study Participants - Enhanced Implementation Arm
Number analyzed (Participants) | 32 | 30
Participants
  Implementation facilitators reported | 16 | 19
  ADMINISTRATION OUTSIDE CLINIC: Home administration by HCP | 24 | 19
  What would do differently | 2 | 4
  Recommended strategies to support patient adherence | 20 | 22

49. Primary Outcome: Number of Participants That Discussed Themes Arising Out of Qualitative Semi-structured Interviews Which Are Coded as Feasibility
Description: A semi-structured interview guide was designed to support the discussion surrounding experience with the implementation of CAB+RPV LA injection treatment. The interview guide topics were informed by the Exploration, Preparation, Implementation, Sustainment (EPIS) framework and Proctor Outcomes to facilitate discussions on the feasibility from the SSPs' perspective. The results of themes that are integral to successful implementation are presented based on implementation strategies.
Time Frame: Up to Month 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Staff Study Participants - Standard Implementation Arm | Staff Study Participants - Enhanced Implementation Arm
Number analyzed (Participants) | 32 | 30
Participants
  No changes made to accommodate clinic needs | 10 | 7
  Changes made to accommodate clinic needs | 22 | 22
  Implementation facilitators reported | 16 | 19
  Developed supplemental materials for implementation | 3 | 5
  Staffing and workload issues was not a challenge | 12 | 7
  Staffing and workload issues was a challenge | 18 | 14
  Staffing and workload issues: How tried to/overcame this challenge | 7 | 10
  Staffing and workload issues: Still a challenge | 7 | 4
  Staffing and workload issues: Not a challenge at present | 8 | 5
  Availability of rooms and designated space: Was not a challenge | 19 | 15
  Availability of rooms and designated space: Was a challenge | 13 | 7
  Availability of rooms and designated space: How overcame this challenge | 9 | 7
  Availability of rooms and designated space: Still a challenge | 8 | 4
  Availability of rooms and designated space: Not a challenge at present | 4 | 3
  Coordination between the clinic and pharmacy: Was not a challenge | 23 | 17
  Coordination between the clinic and pharmacy: Was a challenge | 4 | 9
  Coordination between the clinic and pharmacy: How overcame this challenge | 3 | 6
  Coordination between the clinic and pharmacy: Still a challenge | 3 | 3
  Coordination between the clinic and pharmacy: Not a challenge at present | 0 | 4
  Medication supply and storage: Was not a challenge | 16 | 15
  Medication supply and storage: Was a challenge | 9 | 3
  Medication supply and storage: How tried to/overcame this challenge | 7 | 2
  Medication supply and storage: Still a challenge | 2 | 1
  Medication supply and storage: Not a challenge at present | 5 | 2
  Being able to administer injections: Was not a challenge | 24 | 17
  Being able to administer injections: Was a challenge | 3 | 3
  Being able to administer injections: How overcame this challenge | 1 | 3
  Being able to administer injections: Still a challenge | 1 | 2
  Being able to administer injections: Not a challenge at present | 2 | 1
  Being able to administer injections: ViiV not supportive of CAB+RPV LA implementation | 0 | 5
  Being able to administer injections: ViiV supportive of CAB+RPV LA implementation | 31 | 23
  Being able to administer injections: What would do differently | 2 | 4

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs), non-serious AEs and all-cause mortality were collected up to Month 26.
Description: Adverse events were reported for safety population which comprised of all participants enrolled and who received at least 1 dose of CAB LA+RPV LA. Staff Study Participants (SSP) did not receive oral lead-in medication or CAB+RPV LA injections. Adverse events for SSP were not collected because it was not required per study design.
Arm/Group | Patient Study Participants
All-Cause Mortality (participants affected / at risk) | 0/430
Serious Adverse Events (participants affected / at risk) | 17/430
Other Adverse Events (participants affected / at risk) | 384/430
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Study Participants (N=430)
Appendicitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Yersinia infection (Infections and infestations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Appendicitis noninfective (Gastrointestinal disorders) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Haematospermia (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Orthostatic intolerance (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Varicocele (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Study Participants (N=430)
Injection site pain (General disorders) | 345 (1632)
Injection site induration (General disorders) | 48 (79)
Injection site discomfort (General disorders) | 38 (94)
Pyrexia (General disorders) | 41 (54)
Injection site nodule (General disorders) | 32 (57)
Injection site swelling (General disorders) | 27 (38)
Asthenia (General disorders) | 27 (32)
COVID-19 (Infections and infestations) | 79 (85)
Nasopharyngitis (Infections and infestations) | 30 (33)
Back pain (Musculoskeletal and connective tissue disorders) | 35 (36)
Headache (Nervous system disorders) | 41 (50)
Diarrhoea (Gastrointestinal disorders) | 30 (35)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (26)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT04399551/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT04399551/SAP_002.pdf